CLINICAL TRIAL: NCT04956874
Title: The Florida REACH Translation Project
Brief Title: FL-REACH: Pilot Trial of a Brief Dementia Caregiver Intervention
Acronym: FL-REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Collaborators: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000599
Record Dates: First submitted 2021-06-22; First posted 2021-07-09 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Caregiving; ADRD; Memory Disorders
MeSH Terms: conditions — Alzheimer Disease; Dementia; Memory Disorders

STUDY DESIGN:
Intervention Model Description: Dementia caregivers were recruited initially. When dementia caregiver recruitment was completed, a small control group was recruited.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants will complete the FL-REACH annualized caregiver intervention.
  Interventions: Behavioral: FL-REACH
- Control Group (No Intervention): No-intervention control group

INTERVENTIONS:
Behavioral: FL-REACH — The FL REACH intervention is a 6-session intervention designed to facilitate transition to care following delivery of a memory disorders diagnosis by a MDC team. The intervention focused on an approach that used a toolbox of strategies to tailor skills-based learning, knowledge transmission, and self-care strategies to dementia caregivers. This pilot study focuses on adapting the established REACH II intervention for translation to the clinical setting, with a focus not only on implementation of the key components of the program, but also on feasibility and sustainability. This is part of a stepped-care model that is being developed at the AdventHealth-Orlando MDC. Caregivers of patients will be referred to the FL REACH intervention for foundational training and skills-development.
  Arms: Experimental Group

SUMMARY:
The primary aim of this study is to test feasibility of a modified REACH II intervention in an outpatient clinic.

DETAILED DESCRIPTION:
Primary Aim The primary aim of this study is to test feasibility of a modified REACH II intervention in an outpatient clinic.

Hypothesis:

1. The FL REACH intervention can be implemented reliably in this setting, with fidelity to the model and minimal burden on existing clinic structure.

   Secondary Aims Aim 2: Examine the effectiveness of a REACH II translation in an outpatient setting.

   Hypotheses:
2. CG disease knowledge will increase from pre-assessment to post-assessment.
3. Caregiver preparedness for caregiving will increase from pre-assessment to post-assessment.
4. Perceived risk by CG (CR access to dangerous objects + smoking + supervision + wandering + driving + screaming + desire to hit) will be reduced from pre-assessment to post-assessment.
5. Caregivers will demonstrate mastery of skill acquisition related to behavior change strategies.
6. Caregiver burden will decrease from pre-assessment to post-assessment.
7. Caregiver self-rated health will improve from pre-assessment to post-assessment.
8. Caregivers will have initiated the process of advanced care planning by the end of the intervention.
9. All measures will maintain gain in the anticipated direction from baseline measures at 6 months post-assessment.

Aim 3: Identify possible moderators of outcome, such as race/ethnicity, language, dosage or relationship.

This Aim is exploratory. Based in previous evidence, we estimate similar outcomes for all participants regardless of demographic factors, but previous trials have never been attempted in this novel setting. We will examine the data for differential outcomes related to such factors.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-89 2. Identified caregiver or care partner of an individual who has been diagnosed with Alzheimer's disease or another dementia by the memory disorders clinic, and/or who has sought ongoing treatment through the memory disorders clinic 3. Able to provide informed consent 4. Able to engage in the intervention weekly by attending sessions in person at the clinic 5. Able to participate in the intervention in English or in Spanish 6. No previous experience with a caregiver training program in the past (this applies to theory based, structured interventions delivered by professionals, and does not include peer-led support groups that the family may have engaged with)

Exclusion Criteria:

* 1. Under age of 18 or over the age of 89 2. Unable to provide informed consent or subject to a conflict of interest for this study 3. Unable to return regularly to the clinic for sessions 4. Engaged in another caregiver training program concurrently or have completed a multi-week caregiver training program in the past (this exclusion applies to theory based, structured interventions delivered by professionals, and does not include peer-led support groups that the family may have engaged with)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2020-09-17 (Actual); Study Completion 2020-09-17 (Actual)

PRIMARY OUTCOMES:
Caregiver Burden | Baseline; 6 weeks (therapy termination); 6 month follow-up
  Zarit Burden Inventory
Preparedness for Caregiving Measure | Baseline, session 2, 4, 6 (therapy termination); 6 month follow-up
  Preparedness for dementia caregiving
Alzheimer's disease Knowledge Scale | Baseline, 6 (therapy termination); 6 month follow-up
  Knowledge of Alzheimers Disease and Related Dementias

SECONDARY OUTCOMES:
Risk Assessment | Baseline, 6 (therapy termination); 6 month follow-up
  FL-REACH Risk assessment
FL-REACH Satisfaction Survey | Baseline, 6 (therapy termination); 6 month follow-up
  FL-REACH Satisfaction Survey.
Health Self-Report | Baseline, 6 (therapy termination); 6 month follow-up
  Self-Report of personal health

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - AdventHealth, Orlando, Florida
  - University of Central Florida, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD at this time.